CLINICAL TRIAL: NCT06200623
Title: Cognitive and Emotional Factors Relation to Treatment Adherence in Asthmatic Patients in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Entsar Hsanen (Other)
Responsible Party: Sponsor-Investigator, Entsar Hsanen, Dr, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Cognitive and emotional factor
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Bronchial Asthma; Adherence, Medication
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthmatic patients presented to respiratory outpatient clinic: All subjects will be subjected to Complete history taking including demographic data, residence, educational level, income level, and presence of first- or second-degree medical relative. The first onset age of asthma and duration of asthma will be recorded. Factors that can affect treatment adherence are collected as type and number of medications, cost, inclusion in the health insurance system, availability, asthma-related comorbidities, and choice of drug and device.
  : To assess adherence we will use the Morisky Medication Adherence Scale (MMAS-8) as discussed above
  To assess patient beliefs, we will use The Beliefs about Medicines Questionnaire as discussed above To obtain information on illness perception we will use The Brief Illness Perception Questionnaire (Brief IPQ) as discussed above To assess asthma control we will use the asthma control test as discussed above

SUMMARY:
Non-adherence to controller therapy is one of the main reasons of poor asthma control. Adherence to medication in different studies range between 30 and 70% . Several factors related to the disease, to the patient, treatment or physician- patient relationship

DETAILED DESCRIPTION:
Non-adherence to controller therapy is one of the main reasons for poor asthma control. Adherence to medication in different studies ranges between 30 and 70%. Several factors related to the disease, to the patient, treatment, or physician-patient relationship have been identified to be related to adherence in asthma and other diseases. According to the self-regulation theory, medication beliefs and illness perception are associated with treatment adherence. Beliefs about illness, the necessity, and the concerns (addition and side effects) of the treatment have been identified as the two most important elements in the proposed theory. Other factors that impact treatment adherence are the perceived efficacy of medicines, cost of therapy, complex dosing regimens, Patient's level of education, and cultural beliefs. Evaluating the beliefs about asthma medication, and cognitive and emotional perceptions may help to identify patients with poor adherence to treatment in clinical practice. That would guide additional attention helping to increase the likelihood of taking asthma medication appropriately. However, only limited information is available on treatment adherence in Egyptian people especially in upper Egypt. Furthermore, evidence identifying medication beliefs, and cognitive or emotional factors associated with asthma medication adherence among Egyptian people in upper Egypt is currently not available

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide informed consent.
2. Age ≥18y at the time of study enrollment.
3. Provider diagnosed asthma and prescribed maintenance ICS treatment and as needed bronchodilator for at least one month

Exclusion Criteria:

1. Any other medical condition that confers greater illness morbidity than asthma (e.g., active cancer)
2. Severe psychopathology (e.g., schizophrenia)
3. Apparent cognitive or language deficit
4. Patients with associated other chronic chest diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 138 asthmatic patients presented to respiratory outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence in asthmatic patients in upper Egypt and association to disease beliefs | one year
  simple questionnaires will be used to assess adherence, beliefs, and perception

CONTACTS AND LOCATIONS:
Overall Officials: Entsar H Mohamed, Lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No